CLINICAL TRIAL: NCT04507646
Title: The Effectiveness of Auricular Acupuncture on Improving Secretion of Saliva Among Institutional Older Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Huang, Hui-Chuan, The Effectiveness of Auricular Acupuncture on Improving Secretion of Saliva Among Institutional Older Population, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: N202001048
Record Dates: First submitted 2020-07-26; First posted 2020-08-11 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Salivary Gland Diseases
MeSH Terms: conditions — Salivary Gland Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Two blinded researchers indenpendent performered auricular acupuncture for experimental or control group, respectively.
  Experimental group receive true auricular acupuncture and control group receive sham auricular acupuncture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- True auricular acupuncture (Experimental): Effective auricular acupuncture
  Interventions: Other: True auricular acupuncture
- Sham auricular acupuncture (Sham Comparator): Ineffective auricular acupuncture
  Interventions: Other: sham auricular acupuncture

INTERVENTIONS:
Other: True auricular acupuncture — The participant in experimental group will receive acupuncture on ear Shenmen point, ear zero point, and Salivary glands.
  Arms: True auricular acupuncture
Other: sham auricular acupuncture — The participant in control group will receive acupuncture on ineffective point at ear.
  Arms: Sham auricular acupuncture

SUMMARY:
The study aims to examine the effect of auricular acupuncture on improving oral health in older population. The hypothesis of this study is that older people receiving auricular acupuncture can increase salivary secretion. By identifying the effectiveness of auricular acupuncture can increase salivary secretion; suitable care can be suggested to improve oral health in older population living in long-term institutions.

DETAILED DESCRIPTION:
The elderly living in long-term institutions are mostly limited to physical dysfunction and highly dependence. In addition, the chronic diseases are affected by taking a variety of drugs, which may easily lead to dry mouth. Thus, providing oral health to increase secretion of saliva is high recommended to those older population. The study is used to examine the effect of auricular acupuncture on improving oral health in older population. The eligible participants are random assign to experimental group receiving auricular acupuncture and control group having ineffective auricular acupuncture. Outcome measures include demographic variables, general health status and secretion of saliva, such as: Subjective dry mouth condition and objective mouth condition. Generalized linear model will be used to examine the effect of auricular acupuncture on improving oral health. By identifying the effectiveness of auricular acupuncture can increase salivary secretion; suitable care can be suggested to improve oral health in older population living in long-term institutions.

ELIGIBILITY:
Inclusion Criteria:

1. Residents in long-term institutions aged over 65 years old
2. Living in long-term institutions at least six months and above
3. Having normal cognitive functions with Mini-Mental State Examination scores more than 25 scores.

Exclusion Criteria:

1. The resident whose acupuncture point has Trauma, eczema or ulcer.
2. Incapable of salivary secretion caused by disease,sush as radiation-induced xerostomia among patients with nasopharyngeal carcinoma, Sjogren's Syndrome,acute sialadenitis,chronic recurrent sialadenitis,viral salivary gland infection,salivary gland stones.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Subjective dry mouth health | pre-test and post-test
  self-rated salivation
Objective dry mouth health | pre-test and post-test
  Salivation measured by Oral moisture meter

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chuan Huang, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Yilan Yuanshan Hopsital, Yilan, Taiwan